CLINICAL TRIAL: NCT05751850
Title: HR070803 in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate Versus Nab-paclitaxel in Combination With Gemcitabine for First-line Treatment of Advanced Pancreatic Cancer: an Open, Randomized, Multicenter Phase III Trial.
Brief Title: HR070803 in Combination With Oxaliplatin, 5-FU/LV Versus AG for First-line Treatment of Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR070803-301
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: First-line Treatment of Advanced Pancreatic Cancer
MeSH Terms: interventions — Oxaliplatin; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: HR070803 in combination with oxaliplatin, 5-FU/LV compared with AG
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate (Experimental)
  Interventions: Drug: HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate
- nab-paclitaxel; gemcitabine (Active Comparator)
  Interventions: Drug: nab-paclitaxel; gemcitabine

INTERVENTIONS:
Drug: HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate — HR070803 in combination with oxaliplatin, 5-fluorouracil, calcium folinate
  Arms: HR070803; Oxaliplatin; 5Fluorouracil; Calcium folinate
Drug: nab-paclitaxel; gemcitabine — nab-paclitaxel in combination with gemcitabine
  Arms: nab-paclitaxel; gemcitabine

SUMMARY:
The purpose of this study is to look at the efficacy and safety of HR070803 in combination with 5 fluorouracil/leucovorin (5FU/LV) plus oxaliplatin compared to nab-paclitaxel + gemcitabine treatment in improving the overall survival of patients not previously treated for metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1
2. Histological or cytologically confirmed pancreatic cancer that has not been previously treated in the metastatic disease.
3. Life expectancy of greater than or equal to3 months.
4. At least one measurable lesion is present according to the efficacy evaluation criteria for pancreatic cancer (RECIST 1.1)
5. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Patients with pancreatic cancer originating from extrapancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, acinar cell carcinoma of the pancreas, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Known history of central nervous system (CNS) metastases.
3. Severe infection (> CTCAE grade 2), such as severe pneumonia, bacteremia, infection complications, etc. requiring inpatient treatment, occurred within four weeks before enrollment, and symptoms and signs of infection requiring intravenous antibiotic therapy (except for prophylactic antibiotics) occurred within two weeks before enrollment;
4. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Patients with NYHA class 2 and above cardiac failure; (2) unstable angina; (3) myocardial infarction that occurred within 6 months; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 778 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From study start until 399 OS events have occurred (approximately 15 months after last patient enrollment)

SECONDARY OUTCOMES:
Objective Response rate (ORR) | up to 6 months following the date the last patient was randomized
  ORR is defined as the percentage of participants who have a best overall response of complete response (CR) or partial response (PR), per RECIST 1.1.
Disease Control Rate | up to 6 months following the date the last patient was randomized
  The study is designed to evaluate the disease control rate with advanced pancreatic cancer. DCR is defined as the percentage of patients with a best response of CR, PR, or stable disease (SD).
Duration of Response | up to 6 months following the date the last patient was randomized
  DoR is defined as the time from first documentation of response (CR or PR whichever occurred first, as per RECIST version 1.1) to disease progression or death, whichever is earlier.
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  PFS is defined as the time from the date of first dose of study drug to the date of the first documentation of disease progression or date of death, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided